CLINICAL TRIAL: NCT00323115
Title: A Phase II Feasibility Study of Adjuvant Intra-Nodal Autologous Dendritic Cell Vaccination for Newly Diagnosed Glioblastoma Multiforme
Brief Title: Phase II Feasibility Study of Dendritic Cell Vaccination for Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0536
Record Dates: First submitted 2006-05-04; First posted 2006-05-09 (Estimated); Results first posted 2012-09-26 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Glioblastoma Multiforme
Keywords: immunotherapy; cancer vaccine; glioblastoma multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine (Experimental)
  Interventions: Biological: Autologous Dendritic Cell; Drug: Temozolomide; Procedure: Radiotherapy; Biological: Dendritic Cell Vaccine

INTERVENTIONS:
Biological: Autologous Dendritic Cell — Vaccine given by cervical lymph node injection 3 times every other week
Drug: Temozolomide — Radiotherapy (RT) with concurrent temozolomide (TMZ) for 6 weeks before vaccine is SOC
Procedure: Radiotherapy — RT is standard of care (SOC) post surgery
Biological: Dendritic Cell Vaccine — Vaccine given cervical lymphnode injection 3 times every other week

SUMMARY:
Adult patients who have surgical resection of newly diagnosed glioblastoma multiforme will be treated with radiotherapy/chemotherapy followed by dendritic cell vaccine. Chemotherapy will be administered after three vaccinations for one year or until progression of disease.

DETAILED DESCRIPTION:
Two to six weeks after surgery, patients with newly diagnosed glioblastoma multiforme (GBM) will undergo a six-week course of radiotherapy with concurrent chemotherapy (temozolomide). Between three and seven weeks after completing radiotherapy/chemotherapy, patients will undergo leukapheresis to collect white blood cells. These cells will be grown into dendritic cells, and cultured with tumor cells from the individual patient. Vaccinations will be given every two weeks for a total of three vaccinations. Four weeks after the third vaccination patients will resume chemotherapy for one year or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven GBM with central pathology review at Dartmouth-Hitchcock Medical Center (DHMC)
* Tumor specimen obtained at the time of surgery adequate for vaccination
* 18 years of age or older
* Karnofsky Performance Status 60% or greater
* Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10 9th/L
* Platelets greater than or equal to 100 x 10 9th/L
* Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) less than or equal to 5 times the upper limits of normal (ULN)
* Total bilirubin less than or equal to 1.5 times ULN
* Serum creatinine less than or equal to 1.5 times ULN, OR estimated creatinine clearance greater than or equal to 60 mL/min
* No known immunosuppression other than chemo-related
* Negative HIV serologies
* No evidence of acute or chronic hepatitis on standard hepatitis C and B screening tests
* No chemotherapy within four weeks prior to leukapheresis
* Radiotherapy at outside institution is permitted if tissue was obtained at time of surgery at DHMC and patient is willing to follow-up per protocol
* Off steroids for at least two weeks before leukapheresis
* No second malignancies except non-melanoma skin cancer, and non-invasive cancer such at cervical CIS, superficial bladder cancer or breast CIS
* Negative serum or urine pregnancy test for women of childbearing potential
* No serious uncontrolled medical disorder or active infection
* All patients must give informed consent
* No history of clinical evidence of active autoimmune disease

Exclusion Criteria:

* Invasive cancers in the past 5 years
* Rheumatologic/autoimmune disease
* Pregnancy or unwillingness to remain on acceptable form of birth control during study
* Major cardiac, pulmonary, or other systemic disease; viral hepatitis; HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camilo E. Fadul, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Result] Fadul CE, Fisher JL, Hampton TH, Lallana EC, Li Z, Gui J, Szczepiorkowski ZM, Tosteson TD, Rhodes CH, Wishart HA, Lewis LD, Ernstoff MS. Immune response in patients with newly diagnosed glioblastoma multiforme treated with intranodal autologous tumor lysate-dendritic cell vaccination after radiation chemotherapy. J Immunother. 2011 May;34(4):382-9. doi: 10.1097/CJI.0b013e318215e300. PMID 21499132

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2006 and February 2008, 60 patients were diagnosed with GBM at our institution. Of 11 patients who entered the study, 1 had a seizure with neurologic deterioration several weeks after leukapheresis and did not receive any DC vaccinations.
Groups:
- Vaccine: Adult patients who have surgical resection of newly diagnosed glioblastoma multiforme (GBM) will be treated with radiotherapy and concurrent chemotherapy followed by intranodal vaccine with autologous dendritic cells (DCs) primed with tumor lysate. Adjuvant chemotherapy will be administered after vaccination for 1 year or until tumor progression
Period: Vaccine Administration
Arm/Group | Vaccine
Started | 11
Completed | 10
Not Completed | 1
Not completed — Adverse Event | 1
Period: Adjuvant Therapy & Survival Follow-Up
Arm/Group | Vaccine
Started | 10
Completed | 2
Not Completed | 8
Not completed — Death | 8

BASELINE CHARACTERISTICS:
Arm/Group | Vaccine
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.273 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Tumor-specific Cytotoxic T-cell Response
Description: MRI & pheresis post vaccine
Time Frame: Day 42
Population: All participants who received all 3 vaccine administrations were used in this data analysis.
Measure: Median (Full Range); unit: 10^9 cells/L
Arm/Group | Vaccine
Number analyzed (Participants) | 10
10^9 cells/L
  No. CD4+ | 0.496 [0.198 to 0.921]
  No. CD8+ | 0.4836 [0.135 to 0.976]

2. Secondary Outcome: Number of Adverse Events: Toxicity Profile of Intra-nodal DC/Tumor Lysate Vaccination
Description: Adverse events attributed to vaccination. Collected and attributed adverse events at each study visit; monitored participants for adverse events for two hours following vaccination procedure.
Time Frame: Until death or approximately 24 months after diagnosis
Population: Participants were monitored for adverse events at each visit and observed for 2 hours after intranodal injections. Toxicities were graded using the Common Terminology Criteria for Adverse Events (version 3.0) and Common Toxicity Criteria (version 3.0).
Measure: Number; unit: attributable adverse events
Arm/Group | Vaccine
Number analyzed (Participants) | 10
attributable adverse events | 1

3. Secondary Outcome: Number of Participants With Evaluable Data: Feasibility of Vaccination
Description: To determine the feasibility of this approach, the investigators hypothesize that at least 2/3 of the patients included in the study will be evaluable, meaning that the participants would have received the 3 vaccinations with immunologic outcome parameters measured before and after vaccination. Therefore a maximum of 15 patients would be enrolled in the study to obtain 10 evaluable patients. If after enrolling 15 patients the investigators are unable to obtain 10 evaluable patients, the investigators would consider this approach not feasible.
Time Frame: Through enrollment, approximately 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine
Number analyzed (Participants) | 10
Participants | 10

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival will be assessed for each patient as the time from surgery until the patient reaches objective disease progression by MRI criteria. Death will be regarded as a progression event in those patients that die before disease progression. Patients without documented objective progression at the time of the analysis will be censored at the date of their last objective tumor assessment. Since disease free survival and overall survival are secondary endpoints all patients will be followed until death or for a period of 5 years following enrollment.
Time Frame: Approximately 42 months
Measure: Median (Full Range); unit: Months
Arm/Group | Vaccine
Number analyzed (Participants) | 10
Months | 9.5 [5 to 41]

5. Secondary Outcome: Number of Participants With Significant Difference in Tumor Volume Size Pre- and Postvaccination: Neuroimaging and Tumor Assessment
Description: Patients with evidence of evaluable enhancing disease on contrast-enhanced MRI performed within four weeks of study entry will be evaluated for response rate. Patients will be evaluated for objective tumor assessments by gadolinium-enhanced magnetic resonance imaging (Gd-MRI). Comparisons of objective assessments, excluding progressive disease, are based upon major changes in tumor size on the Gd-MRI compared to the baseline scan. Determination of progressive disease is based upon comparison to the previous scan with volumetric analysis.
Time Frame: baseline and 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine
Number analyzed (Participants) | 10
Participants | 0

6. Secondary Outcome: Overall Survival Duration: Efficacy Parameters
Description: Overall survival will also be followed. Survival will be assessed from the date of surgery to the date of patient death, due to any cause, or to the last date the patient was known to be alive.
Time Frame: Approximately 42 months
Population: There were 4 patients alive when data collection ended, including the patient the longest overall survival.
Measure: Median (Full Range); unit: Months
Arm/Group | Vaccine
Number analyzed (Participants) | 10
Months | 28 [15 to 44]

7. Secondary Outcome: Frequency of CD4+ and CD8+ T Cells - the Proportion of Cells in the Parent Population Responding to Glioblastoma Multiforme (GBM) - Median
Description: Pre- and post-vaccine immune assay results (Tumor-specific T-cells ) are summarized on a continuous scale as median.
Time Frame: Day 7 (pre-vaccination) and Day 42 (post-vaccination).
Population: proportion of cells responding to GBM; GBM = glioblastoma multiforme
Measure: Median (Full Range); unit: proportion of cells
Groups:
- Post-Vaccine: Dendritic Cell Vaccine: Vaccine given cervical lymphnode injection 3 times every other week
Arm/Group | Pre-Vaccine | Post-Vaccine
Number analyzed (Participants) | 10 | 10
proportion of cells
  Precursor frequency of CD4+ T cells | 0.003 [0.0003 to 0.03] | 0.01 [0.0004 to 0.04]
  Precursor frequency of CD8+ T cells | 0.001 [0.0003 to 0.003] | 0.001 [0.0002 to 0.01]

8. Secondary Outcome: Percentage of Tumor-specific T-cells - Correlation Between Immunological Parameters and Efficacy- Median
Description: Pre- and post-vaccine immune assay results (Tumor-specific T-cell Responses) are summarized on a continuous scale as median.
Time Frame: Day 7 (pre-vaccination) and Day 42 (post-vaccination)
Measure: Median (Full Range); unit: percentage of cells
Arm/Group | Pre-Vaccine | Post-Vaccine
Number analyzed (Participants) | 10 | 10
percentage of cells
  Percentage of CD4+ proliferating and IFN | 0.15 [0.004 to 1.96] | 0.25 [0.05 to 5.05]
  Percentage of CD8+ proliferating and IFN | 0.27 [0.01 to 1.45] | 0.25 [0.04 to 4.29]

9. Secondary Outcome: Number of Enzyme-linked Immunosorbent Spots (ELISPOT) - Correlation Between Immunological Parameters and Efficacy - Median
Description: Pre- and post-vaccine immune assay results (Tumor-specific T-cell Responses) are summarized on a continuous scale as mean.
Time Frame: Day 7 (pre-vaccination) and Day 42 (post-vaccination)
Measure: Median (Full Range); unit: spots
Arm/Group | Pre-Vaccine | Post-Vaccine
Number analyzed (Participants) | 10 | 10
spots | 0 [0 to 14] | 0 [0 to 341]

10. Secondary Outcome: Frequency of CD4+ and CD8+ T Cells - the Proportion of Cells in the Parent Population Responding to Glioblastoma Multiforme (GBM) - Mean
Description: Pre- and post-vaccine immune assay results (Tumor-specific T-cells ) are summarized on a continuous scale as mean.
Time Frame: Day 7 (pre-vaccination) and Day 42 (post-vaccination)
Population: proportion of cells responding to GBM; GBM = glioblastoma multiforme
Measure: Mean (Standard Deviation); unit: proportion of cells
Arm/Group | Pre-Vaccine | Post-Vaccine
Number analyzed (Participants) | 10 | 10
proportion of cells
  Precursor frequency of CD4+ T cells | 0.005 (0.009) | 0.01 (0.01)
  Precursor frequency of CD8+ T cells | 0.001 (0.0008) | 0.003 (0.004)

11. Secondary Outcome: Percentage of Tumor-specific T-cells - Correlation Between Immunological Parameters and Efficacy- Mean
Description: Pre- and post-vaccine immune assay results (Tumor-specific T-cell Responses) are summarized on a continuous scale as median. IFN = interferon.
Time Frame: Day 7 (pre-vaccination) and Day 42 (post-vaccination)
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Pre-Vaccine | Post-Vaccine
Number analyzed (Participants) | 10 | 10
percentage of cells
  Percentage of CD4+ proliferating and IFN | 0.38 (0.62) | 0.88 (1.55)
  Percentage of CD8+ proliferating and IFN | 0.45 (0.48) | 0.92 (1.37)

12. Secondary Outcome: Number of Enzyme-linked Immunosorbent Spots (ELISPOT) - Correlation Between Immunological Parameters and Efficacy - Mean
Description: as for outcome 9
Time Frame: Day 7 (pre-vaccination) and Day 42 (post-vaccination)
Measure: Mean (Standard Deviation); unit: spots
Arm/Group | Pre-Vaccine | Post-Vaccine
Number analyzed (Participants) | 10 | 10
spots | 1.40 (4.43) | 44.2 (105.8)

13. Secondary Outcome: Evaluation of T Cell Characteristics
Description: Peripheral blood obtained before starting radiation/ temozolomide (TMZ), and at first and second leukapheresis will be used to do lymphocyte phenotyping. We will determine percentages of CD3+/CD8+/CD45RO+ (memory T-cells), CD3+/CD8+/CD28- (CD8 suppressor T cell phenotype), and CD4+/CD25+ cells at those 3 time points. An anti-human Foxp3 antibody will be used to determine if the CD4+/CD25+ cells are T regulatory cells (TREG) and how the compartmental shift correlates with immunoresponse by other immune parameters as well as to efficacy.
Time Frame: Before starting radiation/Temozolomide and at Day 7 and Day 42.
Measure: Mean (Standard Deviation); unit: percentage of cells
Groups:
- Vaccine - Before Starting Radiation/TMZ; Vaccine - First Leukapheresis; Vaccine - Second Leukapheresis: Adult patients who have surgical resection of newly diagnosed glioblastoma multiforme (GBM) will be treated with radiotherapy and concurrent chemotherapy followed by intranodal vaccine with autologous dendritic cells (DCs) primed with tumor lysate. Adjuvant chemotherapy will be administered after vaccination for 1 year or until tumor progression
Arm/Group | Vaccine - Before Starting Radiation/TMZ | Vaccine - First Leukapheresis | Vaccine - Second Leukapheresis
Number analyzed (Participants) | 10 | 10 | 10
percentage of cells
  % of CD3+/CD8+/CD45RO+ (memory T-cells) | 30.8 (11.2) | 25.8 (9.8) | 19.3 (7.0)
  % CD3+/CD8+/CD28- (CD8 suppressor T cell phenotype | 34.6 (21.0) | 30.5 (18.7) | 23.7 (7.2)
  %CD4+/CD25+ cells | 14.9 (6.8) | 14.1 (5.6) | 11.8 (6.1)
  % of are T regulatory cells (TREG) | 4.0 (2.0) | 3.5 (1.9) | 1.2 (0.7)

14. Secondary Outcome: Immunohistochemistry
Description: Pathologic specimen obtained from patients who require of another surgical resection after vaccination will be examined to determine the characteristics of infiltrating tumor cells.
  Paraffin sections of tumor specimen will be stained by immunohistochemistry with antibodies to identify the components of the inflammatory response. This specimen will be compared to the one obtained at the time of initial surgery and changes in inflammation and inflammatory cellular components will be noted.
Time Frame: Approximately 42 months
Population: Number of patients with pre- and post-tumor tissue procured, to undertake a meaningful analysis of the tumor immunohistochemistry slides inflammatory cells was insufficient. No data was collected.
Arm/Group | Vaccine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Baseline through 30 days after last administration of vaccine.
Description: Participants who started in the "Adjuvant Therapy" Period were assessed for Other/Non-Serious Adverse Events
Arm/Group | Vaccine
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=10)
Pain, neck, unilateral, Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No